CLINICAL TRIAL: NCT04445909
Title: Validation of Continuously Determined Transcutaneous Carbon Dioxide Partial Pressures in Patients Supported with Veno-arterial Extracorporeal Membrane Oxygenation
Brief Title: Validation of Continuous Transcutaneous Carbon Dioxide Monitoring in VA-ECMO Patients
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Martin Dworschak, Assoc. Prof. of Anesthesia and Intensive Care Medicine, Medical University of Vienna
Other Study IDs: 456499
Record Dates: First submitted 2020-05-23; First posted 2020-06-24 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Carbon Dioxide
Keywords: ECMO; Carbon dioxide elimination; Organ perfusion; Low cardiac output; Monitoring; Critical Care
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- VA-ECMO patients: VA-ECMO support because of low cardiac output.
  Interventions: Device: VA-ECMO

INTERVENTIONS:
Device: VA-ECMO — Deployment of extracorporeal membrane oxygenation cardiac assist device.

SUMMARY:
Carbon dioxide in patients on veno-arterial extracorporeal membrane oxygenation (VA-ECMO) is eliminated via respirator as well as via the oxygenator's membrane of the ECMO machine. Consequently, monitoring of end-tidal carbon dioxide tensions is limited, which can result in marked swings towards non-physiological values. Hyper- and hypocapnia, however, can have detrimental effects on organ perfusion in a great number of patients supported with VA-ECMO. Continuous, rapidly applicable monitoring of reliable carbon dioxide measures would therefore be extremely helpful to prevent harmful deviations from the norm. The investigators therefore try to assess the accuracy and the precision of continuously measured non-invasive transcutaneous carbon dioxide partial pressures when compared with tensions determined by blood gas analysis.

DETAILED DESCRIPTION:
After documenting the characteristics of participants, cannulation site, and the cause for ECMO support, transcutaneous, arterial, venous, as well as end-tidal carbon dioxide partial pressure values are measured simultaneously at steady state conditions and compared with each other at various time points over a four-hour observation period. In addition, oxygen tensions are registered transcutaneously and in arterial and venous blood while respirator settings, sweep gas flow, ECMO flow, body temperature, volume status, and the dosage of vasopressors are also being recorded.

ELIGIBILITY:
Inclusion Criteria:

* Low cardiac output requiring VA-ECMO support.

Exclusion Criteria:

* Age < 18 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with low cardiac output after ECMO deployment in tertiary care center.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Agreement between transcutaneous carbon dioxide partial pressure measurement and arterial carbon dioxide partial pressures in VA-ECMO patients. | Through study completion, an average of 2 years
  Bland Altman plot, Pearson correlation, Concordance analysis

SECONDARY OUTCOMES:
Reaction time from attachment of sensor to first reliable reading and its modifiers | Through study completion, an average of 2 years
  Descriptive statistics
Agreement between transcutaneous oxygen partial pressure measurement and arterial oxygen partial pressures in VA-ECMO patients. | Through study completion, an average of 2 years
  Bland Altman plot, Pearson correlation, Concordance analysis
Correlation between transcutaneous carbon dioxide partial pressure level and brain saturation | Through study completion, an average of 2 years
  Pearson correlation, Concordance analysis

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dworschak, MD, MBA, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No